CLINICAL TRIAL: NCT02349672
Title: Clinical Utility of Serum Biomarkers for the Management of Neonatal Hypoxic Ischemic Encephalopathy (HIE) Control Levels
Brief Title: Clinical Utility of Serum Biomarkers for the Management of Neonatal Hypoxic Ischemic Encephalopathy (Control Levels)
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201400671
Record Dates: First submitted 2015-01-23; First posted 2015-01-29 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Hypoxic Ischemic Encephalopathy
Keywords: HIE; Neonates
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control: The healthy control group will have 500-800uL (less than 1 mL) of blood collected. This sample will be obtained at the same time that the neonate is already having a standard blood screenings drawn at 24 and 48 hours of life.
  Interventions: Procedure: blood sample
- Clinical Control: The clinical control group will be healthy neonates that are being evaluated for jaundice, with multiple blood samples drawn between birth and 48 hours of life to monitor serum bilirubin. With these already scheduled lab draws, we will draw an additional 0.8-1 mL of blood.
  Interventions: Procedure: blood sample

INTERVENTIONS:
Procedure: blood sample — Blood will be collected to test for concentrations of UCH-L1 and GFAP.

SUMMARY:
Hypoxic-ischemic encephalopathy (HIE) is a serious birth complication due to systemic asphyxia which occurs in about 20 of 1,000 full-term infants and nearly 60% of premature newborns. Between 10-60% of babies who exhibit HIE die during the newborn period and up to 25% of the HIE survivors have permanent neurodevelopmental handicaps in the form of cerebral palsy, mental retardation, learning disabilities, or epilepsy. HIE also has a significant financial impact on the health care system. In the state of Florida, the total cost for initial hospitalization is $161,000 per HIE patient admitted, but those costs don't take into account the life-long costs.

Current monitoring and evaluation of HIE, outcome prediction, and efficacy of hypothermia treatment rely on a combination of a neurological exam, ultrasound, magnetic resonance imaging (MRI) and electroencephalography (EEG). However, these methods do a poor job in identifying non-responders to hypothermia. MRI requires transport of the neonate with a requisite 40-45 min scan, which is not appropriate for unstable neonates. Moreover, the amplitude integrated EEG (aEEG), a common bedside monitoring technique currently used in these patients to assess candidates and predict outcomes prior to hypothermia, can be adversely affected by hypothermia itself and the patient may not appear to improve until re-warming. Consequently, the development of a simple, inexpensive, non-invasive, rapid biochemical test is essential to identify candidates for therapeutic hypothermia, to distinguish responders from non-responders and to assess outcome. This research is the first step needed to treat neonates with HIE employing a personalized medical approach using serum proteins GFAP and UCH-L1 as biomarkers and by monitoring neonates responses to therapeutic hypothermia. These biomarkers will aid in the direct care by providing a rapid test to predict outcomes and select candidates who are likely to benefit from therapeutic hypothermia and gauge a response to the neuroprotective intervention.

DETAILED DESCRIPTION:
Control Neonates will be easily obtained from a single center, Shands UF. The control samples will be derived from two groups: (1) "Healthy Controls" will be healthy neonates with Apgar scores ≥ 7 at 1 minute and ≥ 8 at 5 minutes and no other medical problems associated with neurologic injury such as hyperbilirubinemia or hypoglycemia. This group will establish a negative control and will have 500-800µL of blood collected at the time of standard blood metabolic screens (at 24 and 48 hours of life). (2) "Clinical Controls" will be healthy neonates evaluated for jaundice, with multiple blood samples drawn between birth and 48 hours of life to monitor serum bilirubin concentrations. They will have an additional 0.8-1 mL of blood drawn at the time of any clinical sample (venous or heel stick) is performed. In addition, neonates will be excluded if they show signs of sepsis or hypoglycemia (< 40). The neonates' bilirubin will be plotted using the American Academy of Pediatrics risk-based stratification method, the Bhutani monogram (which is a based on the serum bilirubin concentration and the hours of life). Clinical control neonates must have low-risk or low-intermediate bilirubin concentrations, with virtually no risk of brain injury.

ELIGIBILITY:
Inclusion Criteria:

* greater than 1.8 kg
* gestational age of 34 weeks or greater

Exclusion Criteria:

* less than 1.8 kg
* gestational age less than 34 weeks

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: neonates
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Levels of UCH-L1 in blood | 72 hours
  Determining if UCH-L1 concentrations measured in neonates with HIE are significantly elevated as compared to controls. Evaluate serum biomarker concentrations from a cohort of neonatal HIE patients who are candidates for hypothermia. These samples will be compared to samples collected from the two cohorts of neonatal "control" subjects.

SECONDARY OUTCOMES:
Levels of GFAP in blood | 72 hours
  Determining if GFAP concentrations measured in neonates with HIE are significantly elevated as compared to controls. Evaluate serum biomarker concentrations from a cohort of neonatal HIE patients who are candidates for hypothermia. These samples will be compared to samples collected from the two cohorts of neonatal "control" subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole R Copenhaver, RN, Study Chair — Study nurse UF Neonatology; Melissa Huene, RN, Study Chair — Study nurse UF Neonatology
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided